CLINICAL TRIAL: NCT07228533
Title: Evaluation of the Effectiveness of a Nursing-Based Co-Design Intervention Program (CesiKids) to Enhance Psychological Resilience in Hospitalized Adolescents Diagnosed With Cancer: A Randomized Controlled Trial
Brief Title: CesiKids Trial: Enhancing Psychological Resilience in Adolescents With Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Sibel Dağliyar, PhD Candidate, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ESOGU-SBF-SD-01
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Resilience, Psychological; Adolescent Cancer; Mobile Application; Pediatric Cancer; Pediatric Nursing; Coping
Keywords: Adolescent; Resilience; Coping skills; Neoplasms; Pediatric nursing; Mobile application; Psychosocial intervention
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial with a parallel assignment design. Participants will be randomly assigned to either the intervention or control group and followed concurrently. Adolescents in the intervention group will participate in the four-week CesiKids mobile psychosocial resilience program, while the control group will receive standard clinical care. No crossover between groups will occur.
Who Masked: Outcomes Assessor
Masking Description: Since the study will be conducted by the principal investigator, investigator blinding will not be possible. Additionally, because the study will be carried out with hospitalized adolescents and the intervention and control groups will be present in the clinic simultaneously, participant blinding cannot be implemented. To prevent potential bias in group allocation, the randomization table will be generated by an independent statistician. Data analysis and reporting will also be conducted by the same independent statistician, ensuring blinding at the statistical analysis stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Psychosocial Care Group (No Intervention): Participants in this arm will receive standard psychological care routinely provided within the pediatric oncology clinic. No additional structured digital intervention or psychological resilience-based program will be administered. Standard support, including routine clinical communication and psychological services offered by the healthcare team, will continue as usual during the study period.
- CesiKids Intervention Group (Experimental): Participants in this group will receive the CesiKids program, a mobile-based psychological resilience intervention specifically developed for adolescents diagnosed with cancer. The program includes AI-supported guidance and interventions and consists of a total of four modules delivered over four weeks, with two structured sessions per module (eight sessions in total). Participants' engagement with the program and their assessment outcomes will be evaluated to determine the feasibility and effectiveness of the CesiKids intervention in enhancing psychological resilience and coping skills among adolescents with cancer.
  Interventions: Other: CesiKids Mobile-Based Psychological Resilience Program

INTERVENTIONS:
Other: CesiKids Mobile-Based Psychological Resilience Program — The CesiKids Program will be a nurse-led, AI-supported mobile intervention to enhance psychological resilience in adolescents diagnosed with cancer. Grounded in Bronfenbrenner's Bioecological Theory, it will address interactions between adolescents and their family, peers, and clinical environments. Developed through a co-design process with nurses, recovered adolescents, and parents, the program will include AI-driven adaptive feedback and emotional support features. Delivered over four weeks with structured digital sessions, CesiKids will promote emotional regulation, coping, and resilience through interactive storytelling, reflection, and personalized guidance. This integrative model will combine ecological principles, AI personalization, and participatory design to create an innovative psychosocial care approach for hospitalized adolescents with cancer.
  Other Names: CesiKids Psychological Resilience Intervention; CesiKids Mobile Application; CesiKids Program
  Arms: CesiKids Intervention Group

SUMMARY:
This study will develop and evaluate a mobile-based co-design intervention (CesiKids) to enhance psychosocial resilience in hospitalized adolescents aged 12-18 diagnosed with cancer. The program will be created using Bronfenbrenner's Ecological Systems Theory and designed in collaboration with nurses, recovered adolescents, and parents. A randomized controlled design will be used. The intervention group will participate in a four-week structured program, while the control group will receive standard care. Psychosocial resilience and coping outcomes will be assessed at baseline, post-intervention, and follow-up. This research aims to offer an evidence-based, scalable model to support resilience among adolescents with cancer in clinical settings.

DETAILED DESCRIPTION:
This study aims to develop an innovative mobile-based co-design intervention program to strengthen psychosocial resilience among adolescents aged 12-18 diagnosed with cancer. The program will be structured based on Bronfenbrenner's Ecological Systems Theory, addressing adolescents' individual characteristics, family and close-social environment, and broader ecological interactions in a holistic manner. To date, no study has implemented a theoretically grounded, mobile psychosocial intervention designed specifically to enhance resilience in adolescents with cancer through a co-design process involving nurses, recovered adolescents, and parents. This project aims to fill this gap by presenting a model that can be integrated into both clinical practice and educational settings.

The research will be conducted using a randomized controlled experimental design with intervention and control groups. The intervention group will participate in the newly developed mobile CesiKids program and engage in structured sessions for four weeks to enhance psychosocial resilience skills. The control group will receive standard clinical care. Participants' coping and psychosocial resilience levels will be measured using the Pediatric Cancer Coping Scale (PCCS) and the Child and Youth Resilience Measure (CYRM-R). Data collection will take place at baseline (T0), post-intervention (T1) and during follow-up assessments (T2 and T3). Quantitative data will be analyzed statistically, and the feasibility and usability of the program will also be monitored.

The CesiKids application will be developed by the project leader and research team. Data collection will be carried out by a nurse researcher experienced in pediatric oncology. All intervention, data collection, and analysis procedures will be carefully planned and monitored. All study data will be anonymized and accessible only to the research team. Data will be securely stored on protected servers and maintained throughout the project. All research processes will be conducted in accordance with ethical standards, and participant rights will be fully respected.

The project is expected to generate an evidence-based model that enhances psychosocial resilience among adolescents with cancer. The developed program will be applicable and scalable in both clinical and educational environments. Findings will be disseminated through academic publications, conference presentations, and among relevant healthcare institutions to ensure sustainability and maximize societal impact. Ultimately, this study intends to provide a practical contribution to the field of adolescent psychosocial resilience and to support the adaptation of similar interventions for other chronic illness groups.

ELIGIBILITY:
Inclusion Criteria:

* Parents have provided informed consent after receiving information,
* The child has given assent to participate after being informed,
* The child is between 12 and 18 years of age,
* The child has been diagnosed with cancer and is currently receiving inpatient treatment,
* The child is undergoing chemotherapy and/or radiotherapy,
* The child is able to use a computer and/or smartphone,
* The child can understand and speak Turkish.

Exclusion Criteria:

* Receiving hematopoietic stem cell transplantation treatment,
* Having developed a relapse after remission,
* Experiencing communication difficulties (e.g., intellectual disability, visual impairment, etc.),
* Having a psychiatric diagnosis made by a psychiatrist,
* Having experienced a significant life event affecting psychological well-being within the past four weeks (e.g., death, divorce, etc.).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Child and Youth Resilience Measure (CYRM-R) | Baseline (prior to intervention), immediately post-intervention (within 1 week after completion), 3 months post-intervention, and 6 months post-intervention
  The Child and Youth Resilience Measure-Revised (CYRM-R) is a multidimensional scale based on the socio-ecological model to assess resilience. The 28-item original version was developed by Liebenberg, Ungar, and Van de Vijver through the International Resilience Project. Later, Liebenberg, Ungar, and LeBlanc created a 12-item short form with three subscales: individual, relational, and contextual resilience. Factor loadings ranged from .39-.88, and Cronbach's alpha was .84. Items are rated on a five-point Likert scale (1-5), with higher scores indicating greater resilience. The Turkish adaptation by Arslan showed strong reliability (α = .91; item-total correlations = .45-.79). In this study, the CYRM-R will assess changes in adolescents' resilience after the CesiKids program.

SECONDARY OUTCOMES:
Pediatric Cancer Coping Scale (PCCS) | Baseline (prior to intervention), immediately post-intervention (within 1 week after completion), 3 months post-intervention, and 6 months post-intervention
  The scale was developed by Wu et al. to assess coping strategies among adolescents aged 7-18 diagnosed with cancer. The Turkish validity and reliability study was conducted by Şengül and Törüner with children in the same age range. The scale includes 33 items across three dimensions: cognitive coping, problem-focused coping, and defensive coping. Items are rated on a 0-3 scale, with total scores ranging from 0 to 99. Higher scores indicate stronger coping strategies. The original version showed a Cronbach's alpha of 0.91, while the Turkish version reported 0.77. The scale has been used to assess coping levels in pediatric oncology populations. In this study, it will be used to evaluate the effectiveness of the CesiKids program in enhancing adolescents' coping skills with cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Ayfer AÇIKGÖZ, PhD, Study Director — Eskişehir Osmangazi University Faculty of Health Sciences
Locations (1):
- Ankara University Faculty of Medicine Cebeci Research and Practice Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy and confidentiality concerns. The dataset contains sensitive clinical and psychological information of adolescent patients with cancer, and data sharing could risk participant identification. Only aggregated and anonymized results will be reported in publications.